CLINICAL TRIAL: NCT06456190
Title: Testing STAR and TextSTAR: A Video and Text Messaging Intervention for Recent Sexual Violence Survivors
Brief Title: Testing STAR and TexSTAR: A Video and Text Messaging Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0299; 1R61DA059897-01 (NIH); A487400 (Other: UW Madison); L&S/PSYCHOLOGY/PSYCHOLOGY (Other: UW Madison); Protocol Version 8/28/2025 (Other: UW Madison)
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Sexual Violence; Posttraumatic Stress Disorder; Opioid Use; Opioid Misuse
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Opioid-Related Disorders | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Video, Above Threshold, Text (Experimental): Participants in this condition will receive the STAR intervention video and those who are above threshold on PTSD or opioid misuse at 1 week will be randomized to receive the textSTAR intervention.
  Interventions: Behavioral: Skills Training in Active Recovery (STAR) Video; Behavioral: Text Skills Training in Active Recovery (TextSTAR) program
- Video, Above Threshold, No Text (Experimental): Participants in this condition will receive the STAR intervention video and those who are above threshold on PTSD or opioid misuse at 1 week will be randomized to not receive textSTAR.
  Interventions: Behavioral: Skills Training in Active Recovery (STAR) Video
- Video, Below Threshold (Experimental): Participants in this condition will receive the STAR intervention video and will be below threshold on PTSD and opioid misuse at 1 week and will not be randomized to receive further intervention.
  Interventions: Behavioral: Skills Training in Active Recovery (STAR) Video
- No Video, Above Threshold, Text (Experimental): Participants in this condition will not receive the STAR intervention video and those who are above threshold on PTSD or opioid misuse at 1 week will be randomized to receive the textSTAR intervention.
  Interventions: Behavioral: Text Skills Training in Active Recovery (TextSTAR) program
- No Video, Above Threshold, No Text (No Intervention): Participants in this condition will not receive the STAR intervention video and those who are above threshold on PTSD or opioid misuse at 1 week will not be randomized to receive the textSTAR intervention.
- No Video, Below Threshold (No Intervention): Participants in this condition will not receive the STAR intervention video and will be below threshold on PTSD and opioid misuse at 1 week and will not be randomized to receive further intervention.

INTERVENTIONS:
Behavioral: Skills Training in Active Recovery (STAR) Video — a 12-15 minute video that includes psychoeducation about ptsd and substance misuse plus tips to not avoid safe but scary situations, cope with distress and urges to use, and engage with social support to aid recovery
  Arms: Video, Above Threshold, No Text; Video, Above Threshold, Text; Video, Below Threshold
Behavioral: Text Skills Training in Active Recovery (TextSTAR) program — a 3-week daily text program that includes supportive/empowering messages along with brief coping tips to not avoid safe but scary situations, cope with distress and urges to use, and engage with social support to aid recovery
  Arms: No Video, Above Threshold, Text; Video, Above Threshold, Text

SUMMARY:
This NIDA-funded HEAL Initiative: Opioid Use Disorder Care Pathways for Individuals with Histories of Exposure to Violence R61 seeks to develop and test a brief video intervention to deliver during Sexual Assault Nurse Examiner (SANE) care and a brief text messaging intervention to deliver in the month after the assault to prevent the onset or escalation of PTSD and opioid misuse among survivors of sexual assault.

DETAILED DESCRIPTION:
This pilot trial is part of a larger R61/R33 to test the effectiveness of brief video and text messaging interventions on PTSD and opioid misuse among recent survivors of sexual assault presenting for medical care. In the R61 phase, researchers are working with a sexual assault advisory board to develop the video and text interventions. The research team is partnering with 5-6 Sexual Assault Nurse Examiner programs across the United States to recruit 50 participants. In this pilot trial, researchers aim to test the feasibility of recruitment strategies, acceptability of the interventions among survivors, and preliminary effectiveness of the interventions at addressing PTSD and opioid misuse.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 or older
* Can read and respond to questions in English
* Are receiving a SANE exam for sexual assault victimization within the previous week (7 days)
* Not currently or about to be hospitalized for severe injuries, suicidality, or psychosis
* Not currently or about to be incarcerated

Exclusion Criteria:

* Patients under age 18
* Those who cannot read and respond to questionnaires in English
* Those seeking care that does not include a SANE exam
* Those who cannot consent to receive SANE care.
* Those who are currently or about to be hospitalized for severe injuries, suicidality, or psychosis
* Those who are currently or about to be incarcerated (e.g., suspects, those who have experienced sexual assault within a prison setting and are returning to that setting, etc)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women and nonbinary sexual assault survivors will be invited to participate
Enrollment: 50 (Actual)
Dates: Start 2025-03-12 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Change in Opioid Misuse | 1 week to 1 month
  Assessed using Tobacco, Alcohol, Prescription Medication, and Other Substance (TAPS) Tool.
  The TAPS tool is a brief, two-part assessment of substance use and misuse. The TAPS-1 is a screener with 4 items assessing frequency of use of tobacco, alcohol, prescription medication, and illicit substances. Any response other than "never" on the TAPS-1 indicates a positive screen, which leads to administration of the TAPS-2. The TAPS-2 is a brief assessment including 3-4 yes/no questions for each class of substances assessing level of use, dependence, and concern from others. Cut-offs for problematic substance use and substance use disorder are based on scores on the TAPS-2.
Change in Posttraumatic Stress Disorder | 1 week to 1 month
  Assessed using PTSD Checklist for DSM-5 (PCL-5). The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Scores range from 0-80, with scores of 31 or higher indicating probable PTSD.

SECONDARY OUTCOMES:
Tobacco, Alcohol, and Other Drug Use | 1 month
  Tobacco, Alcohol, Prescription Medication, and Other Substance (TAPS) Tool. The TAPS-1 is a screener with 4 items assessing frequency of use of tobacco, alcohol, prescription medication, and illicit substances. Any response other than "never" on the TAPS-1 indicates a positive screen, which leads to administration of the TAPS-2. The TAPS-2 is a brief assessment including 3-4 yes/no questions for each class of substances assessing level of use, dependence, and concern from others. Cut-offs for problematic substance use and substance use disorder are based on scores on the TAPS-2.
Opioid misuse severity | 1 month
  Assessed using Current Opioid Misuse Measure (COMM), which is a brief patient self-assessment to monitor chronic pain patients on opioid therapy. It is a 17-item questionnaire with a 0-4 point Likert scale. Scores range from 0-68, with higher scores (above 9) indicating the participant may be exhibiting aberrant behaviors associated with misuse of opioid medications.
Depression level | 1 month
  Assessed using the Patient Health Questionnaire-9 (PHQ-9) The PHQ-9 is an 9-item questionnaire where participants report how often in the past 2 weeks they were bothered by specific problems. It is scored on a 4-point Likert scale where 0 = not at all to 3 = nearly every day. The total possible range of scores is 0-27 where higher scores indicate more depressive symptoms.
Mindfulness skills usage | 1 week, 2 week, 3 week, 1 month
  Assessed with 10 items from the Dialectical Behavior Therapy (DBT) skills subscale of the Ways of Coping Checklist, a 38 item self-report instrument that assesses DBT skills utilization in the past week on a scale from 0 = never to 3 = regularly. The checklist has excellent psychometric properties and has been shown to discriminate patients who received skills training during treatment from those who did not. Higher scores reflect greater skills utilization.
Perceived control over recovery process | 1 month
  Assessed with the 8-item Perceived Present Control subscale of the Perceived Control Over Stressful Events Scale. The scale has excellent psychometric properties and higher scores (which reflect greater perceived control) have been associated with recovery following sexual violence.
Opioid craving | 1 week, 2 week, 3 week, 1 month
  Assessed with the Opioid Craving Visual Analog Scale which ranges from 0 = No Craving At All to 100 = Strongest Craving Ever.
Pain severity | 1 week, 2 week, 3 week, 1 month
  Assessed with the Brief Pain Inventory (BPI), a 4-item self-report measure that asks participants to rate their worst pain in the last week, their least pain in the last week, their pain on average, and their pain right now on a scale from 0 = no pain at all to 10 = pain as bad as you can imagine. An overall pain severity score is computed by taking the mean of the four items.
Alcohol use severity | 1 month
  Assessed with the 10-item Alcohol Use Disorders Identification Test (AUDIT), which quantifies consequences or problems associated with alcohol use. Scores of 8 or higher on the AUDIT indicate substantial alcohol problems.
Drug use severity | 1 month
  Assessed with the 10-item Drug Abuse Screening Test (DAST-10), which quantifies consequences or problems associated with drug use. Scores of 6 or higher or the DAST-10 indicate substantial drug use problems.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Walsh, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No